CLINICAL TRIAL: NCT03040050
Title: Rapid PCR to Guide Antibiotic Therapy at the Time of Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 16-386
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Antibiotic Therapy; Prostate Biopsy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The rPCR results will be provided to the clinical provider for the Interventional group participants. The rPCR results will not be provided to the clinic provider for the control group participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men scheduled for prostate biopsy randomized to Control (Other)
  Interventions: Other: Control group
- Men scheduled for a prostate biopsy randomized to Intervention (Experimental)
  Interventions: Other: rPCR results

INTERVENTIONS:
Other: rPCR results — Interventional group: rPCR results will be shared with the clinical provider to determine appropriate standard of care antibiotic treatment at time of standard of care prostate biopsy.
  Arms: Men scheduled for a prostate biopsy randomized to Intervention
Other: Control group — Control group: rPCR results will not be shared with the clinical provider at time of standard of care prostate biopsy. Standard of care antibiotic selection will be up to the discretion of the clinical provider.
  Arms: Men scheduled for prostate biopsy randomized to Control

SUMMARY:
The study is a randomized controlled trial. Subjects are randomly assigned 1:1 to receive either rapid multiplex qPCR (intervention) prior to standard of care prostate biopsy or standard of care (control) prostate biopsy. The subjects will have a rectal culture swab performed prior to the prostate biopsy. One rectal culture swab will be used for rapid multiplex qPCR and the other swab will be sent to microbiology for a standard culture. The subjects randomized to the intervention group will have the qPCR results shared with the physician to determine if additional standard of care antibiotics are needed at time of standard of care prostate biopsy. The subjects randomized to the control group will not have the qPCR results shared with the physician to determine if additional standard of care antibiotics are needed at time of standard of care prostate biopsy. Approximately, 10 days after the prostate biopsy, the research staff will conduct a chart review and/or telephone call to ask about any prostate biopsy infections and complications.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give informed consent
* Be age 50 or older
* Recommended to undergo a prostate biopsy
* No allergy or side effect to fluoroquinolone antibiotics
* No history of prostate biopsy infection
* No hepatic or renal insufficiency in which fluoroquinolone antibiotics are contraindicated.

Exclusion Criteria:

* Unable to give informed consent
* Age < 50
* Not recommended to have prostate biopsy
* Allergic to or have side effects to fluoroquinolone antibiotics
* History of prostate biopsy infection
* Hepatic or renal insufficiency in which fluoroquinolones antibiotics are contraindicated.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Results of rapid qPCR to determine standard of care antibiotic prophylaxis for prostate biopsy. | Day of prostate biopsy
  Reduction in dual antibiotic prophylaxis in the intervention vs.usual care groups.

SECONDARY OUTCOMES:
Determine if rapid qPCR test results in longer patient wait times. | Day of prostate biopsy
  Difference in the amount of time the PCR technique takes compared to the fastest workflow (physician chooses no additional antibiotics).
Determine if rPCR results and standard rectal culture results are the same. | 1 week
  Comparison of rPCR results to standard rectal culture on Fluoroquinolone infused MacConkey agar.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Liss, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- South Texas Veterans Health Care, San Antonio, Texas, United States